CLINICAL TRIAL: NCT06598098
Title: MAMA Tot - Healthy Weight Parallel Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Linda May, Associate Professor; Dept. Chair, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20-002367
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pregnancy Related
Keywords: exercise modes; exercise intervention

STUDY DESIGN:
Intervention Model Description: Pregnant women will be randomized to one of four groups: aerobic exercise, resistance exercise, combination (aerobic + resistance), or control (no exercise). All exercise participants will be prescribed exercise that meets guidelines of the American College of Obstetricians and Gynecologists (ACOG), American College of Sports Medicine (ACSM), and the American Heart Association (AHA); 150 minutes per week, moderate intensity (60-80% aerobic capacity, Rating of Perceived Exertion, rating of perceived exertion (RPE), 12-15) per week. These limits are the same as those that generated previous positive findings for our preliminary data.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Aerobic Exercise (AE) (Experimental): All exercise participants will be prescribed exercise that meets guidelines of the American College of Obstetricians and Gynecologists (ACOG), American College of Sports Medicine (ACSM), and the American Heart Association (AHA); 150 minutes per week, moderate intensity (60-80% aerobic capacity, Rating of Perceived Exertion, RPE, 12-15) per week. These limits are the same as those that generated previous positive findings for our preliminary data. The AE group will exercise on aerobic machines (i.e. treadmill, elliptical, bicycle) for all of their sessions.
  Interventions: Behavioral: Exercise Modes
- Resistance Exercise (RE) (Experimental): All exercise participants will be prescribed exercise that meets guidelines of the American College of Obstetricians and Gynecologists (ACOG), American College of Sports Medicine (ACSM), and the American Heart Association (AHA); 150 minutes per week, moderate intensity (60-80% aerobic capacity, Rating of Perceived Exertion, RPE, 12-15) per week. These limits are the same as those that generated previous positive findings for our preliminary data. The RE group will perform 12-15 repetitions of 10-12 resistance exercises in a circuit, for 3 sets with rest period of 30-60 seconds between sets as needed.[100] Seated isokinetic exercise using Cybex machines will target all major muscle groups. Light dumbbells and resistance bands will be used if the participant is unable to lift the minimal load on Cybex machines. Core exercises will be performed at the end of the session (i.e. seated side bends).
  Interventions: Behavioral: Exercise Modes
- Combination Exercise (AERE) (Experimental): All exercise participants will be prescribed exercise that meets guidelines of the American College of Obstetricians and Gynecologists (ACOG), American College of Sports Medicine (ACSM), and the American Heart Association (AHA); 150 minutes per week, moderate intensity (60-80% aerobic capacity, Rating of Perceived Exertion, RPE, 12-15) per week. These limits are the same as those that generated previous positive findings for our preliminary data. The AERE group will switch between AE exercise and RE; for this group, RE exercises will consist of 1 set of 12-15 repetitions of 4 resistance exercises, then 5 minutes of AE, then repeated repeat with different exercises.[106-108] The investigators will also calculate the metabolic minutes per week (METmin/wk) of all participants in order to account for potential differences in energy expenditure based on activity, though the dose of 150 min/wk at moderate intensity is held constant between exercise groups.
  Interventions: Behavioral: Exercise Modes
- Control (no exercise) (No Intervention): The Control group will participate in weekly sessions that focus on stretching, breathing, and healthy lifestyle.

INTERVENTIONS:
Behavioral: Exercise Modes — Moderate intensity aerobic exercise, moderate intensity resistance exercise, moderate intensity combination exercise
  Arms: Aerobic Exercise (AE); Combination Exercise (AERE); Resistance Exercise (RE)

SUMMARY:
The overall objective of this proposal is to conduct a longitudinal prospective study of healthy pregnant women and their offspring to determine which antenatal maternal exercise mode(s) will have the greatest impact on maternal and infant cardiometabolic health. This information may lead to modified clinical practice recommendations that improve health in childhood and possibly beyond. This randomized controlled trial will recruit 268 healthy pregnant women randomized to an exercise intervention (aerobic exercise, resistance exercise, aerobic and resistance exercise) or to no exercise (usual care); their infants will be measured at 1, 6, and 12 months of age. This rigorous design will test our central hypothesis that aerobic and resistance exercise and resistance exercise training during pregnancy will, in healthy weight BMI (HW) women, improve maternal and offspring cardiometabolic outcomes to a greater extent than AE alone. We will test this hypothesis with two specific aims:

Aim 1. Determine the influence of different exercise modes during HW pregnancy on infant cardiometabolic health and growth trajectories. Hypothesis: AE, RE, and AERE by HW pregnant women will improve offspring neuromotor and cardiometabolic measures at 1, 6, and 12 months postpartum (e.g. decreased % body fat, BMI z-score, heart rate, non-HDL, and C-Reactive Protein (CRP); increased insulin sensitivity) compared to infants of HW pregnant women that do not exercise; AERE and RE will have the greatest impact on improving infant measures.

Aim 2. Determine the most effective exercise mode in HW pregnancy on improving maternal cardiometabolic health outcomes. Hypothesis: AE, RE, and AERE by HW pregnant women will improve both maternal cardiometabolic health measures (e.g. decreased BMI z-score, non-HDL, % body fat, HR, weight gain) across pregnancy (16 to 36 weeks gestation) and overall pregnancy outcomes (e.g. lower incidence of gestational diabetes, pre-eclampsia, hypertension during gestation) compared to HW pregnant women that do not exercise; AERE and RE will have the greatest impact on improving maternal health measures, with the AERE group having the highest compliance.

The proposed innovative study will be the first to provide a critical understanding of the influence of antenatal exercise modes upon the cardiometabolic health and growth trajectories of offspring who may be at increased risk of poor outcomes. This work will have a significant impact on reducing the cycle of OB and CVD, potentially providing the earliest and most efficacious intervention to attenuate or prevent OB and CVD in the next generation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 40 years old
* BMI 18.5 to 24.4
* Pregnancy: Singleton; ≤ 16 weeks gestation
* Clearance by Obstetric provider for exercise

Exclusion Criteria:

* Age: ≤ 17.9 or ≥ 41 years of age
* BMI ≥25
* Multi fetal pregnancy
* Obstetric Provider does not provide clearance for exercise
* Unable or Unwilling to provide consent
* Inability to communicate with members of study team, despite use of interpreter
* Medical Conditions (e,g. HIV/Aids, Cancer, Type 1 or 2 Diabetes, Untreated Hypertension, Thyroid Disorders)
* Use of tobacco products, alcohol, recreational drugs, or medications (oral hypertensive, insulin)
* Unable to provide phone or email contact

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 268 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
1 month Infant non-HDL | 1 month
  non-HDL measures from venipuncture
6 month Infant non-HDL | 6 months
  non-HDL measures from venipuncture
12 month Infant non-HDL | 12 months
  non-HDL measures from venipuncture
1 month infant BMI z-score | 1 month
  BMI normalized
6 month infant BMI z-score | 6 months
  BMI normalized
12 month infant BMI z-score | 12 months
  BMI normalized
Enrollment (8-13wks) Maternal fasting non-HDL | enrollment (~8-13 wks gestation)
  non-HDL measured from venipuncture
36wk Maternal fasting non-HDL | 36wks gestation
  non-HDL measured from venipuncture
1 month Maternal fasting non-HDL | 1 month postpartum
  non-HDL measured from venipuncture
6 month Maternal fasting non-HDL | 6 months postpartum
  non-HDL measured from venipuncture
Adverse Pregnancy Outcomes | At delivery
  Presence or absence of Adverse Pregnancy outcomes (preterm birth, gestational diabetes [GDM], preeclampsia, hypertension)
12 month Maternal fasting non-HDL | 12 months postpartum
  non-HDL measured from venipuncture

SECONDARY OUTCOMES:
1 month infant Resting Heart Rate | 1 month
  resting HR
6 month infant Resting Heart Rate | 6 months
  resting HR
12 month infant Resting Heart Rate | 12 months
  resting HR
1 month infant Resting Blood Pressure | 1 month
  resting BP
6 month infant Resting Blood Pressure | 6 months
  resting BP
12 month infant Resting Blood Pressure | 12 months
  resting BP
1 month infant Body Fat % | 1 month
  body fat % from skinfolds
6 month infant Body Fat % | 6 months
  body fat % from skinfolds
12 month infant Body Fat % | 12 months
  body fat % from skinfolds
1 month infant % Muscle Mass | 1 month
  muscle mass % from skinfolds
6 month infant % Muscle Mass | 6 months
  muscle mass % from skinfolds
12 month infant % Muscle Mass | 12 months
  muscle mass % from skinfolds
1 month Infant Resting Energy Expenditure (REE) | 1 month
  resting REE
6 month Infant Resting Energy Expenditure (REE) | 6 months
  resting REE
12 month Infant Resting Energy Expenditure (REE) | 12 months
  resting REE
1 month Infant Neuromotor Assessment | 1 month
  Peabody Developmental Motor Scale (1st - 99th percentile) - the higher the percentile the better
6 month Infant Neuromotor Assessment | 6 months
  Peabody Developmental Motor Scale (1st - 99th percentile) - the higher the percentile the better
12 month Infant Neuromotor Assessment | 12 months
  Peabody Developmental Motor Scale (1st - 99th percentile) - the higher the percentile the better
1 month Infant Veggie Meter | 1 month
  Raman Spectroscopy-Skin Carotenoid assessments
6 month Infant Veggie Meter | 6 months
  Raman Spectroscopy-Skin Carotenoid assessments
12 month Infant Veggie Meter | 12 months
  Raman Spectroscopy-Skin Carotenoid assessments
1 month Infant Blood Biomarkers (CRP) | 1 month
  Multiplex analyses of inflammatory markers (CRP)
6 month Infant Blood Biomarkers (CRP) | 6 months
  Multiplex analyses of inflammatory markers (CRP)
12 month Infant Blood Biomarkers (CRP) | 12 months
  Multiplex analyses of inflammatory markers (CRP)
1 month Infant Blood Biomarkers (IL6) | 1 month
  Multiplex analyses of inflammatory markers (IL6)
6 month Infant Blood Biomarkers (IL6) | 6 months
  Multiplex analyses of inflammatory markers (IL6)
12 month Infant Blood Biomarkers (IL6) | 12 months
  Multiplex analyses of inflammatory markers (IL6)
1 month Infant Blood Biomarkers (adiponectin) | 1 month
  Multiplex analyses of inflammatory markers (adiponectin)
6 month Infant Blood Biomarkers (adiponectin) | 6 months
  Multiplex analyses of inflammatory markers (adiponectin)
12 month Infant Blood Biomarkers (adiponectin) | 12 months
  Multiplex analyses of inflammatory markers (adiponectin)
1 month Infant Metabolomics | 1 month
  Metabolomic pathway analysis of significantly different blood metabolites based on p-value less than or equal to 0.05
6 month Infant Metabolomics | 6 months
  Metabolomic pathway analysis of significantly different blood metabolites based on p-value less than or equal to 0.05
12 month Infant Metabolomics | 12 months
  Metabolomic pathway analysis of significantly different blood metabolites based on p-value less than or equal to 0.05
16wk Maternal Resting Heart Rate | 16wks gestation
  resting HR
36wk Maternal Resting Heart Rate | 36wks gestation
  resting HR
1 month Postpartum Maternal Resting Heart Rate | 1 month postpartum
  resting HR
6 month Postpartum Maternal Resting Heart Rate | 6 months postpartum
  resting HR
12 month Postpartum Maternal Resting Heart Rate | 12 months postpartum
  resting HR
16wk Maternal Resting Blood Pressure | 16wks gestation
  resting BP
36wk Maternal Resting Blood Pressure | 36wks gestation
  resting BP
1 month Postpartum Maternal Resting Blood Pressure | 1 month postpartum
  resting BP
6 month Postpartum Maternal Resting Blood Pressure | 6 months postpartum
  resting BP
12 month Postpartum Maternal Resting Blood Pressure | 12 months postpartum
  resting BP
Maternal Gestational Weight Gain (GWG) | At delivery
  Gestational Weight Gain
16wk Maternal Body Fat % | 16wks gestation
  estimated body fat %
36wk Maternal Body Fat % | 36wks gestation
  estimated body fat %
1 month Postpartum Maternal Body Fat % | 1 month postpartum
  estimated body fat %
6 month Postpartum Maternal Body Fat % | 6 months postpartum
  estimated body fat %
12 month Postpartum Maternal Body Fat % | 12 months postpartum
  estimated body fat %
16wk Maternal Biomarkers (CRP) | 16wks gestation
  Multiplex analyses of inflammatory markers (CRP)
36wk Maternal Biomarkers (CRP) | 36wks gestation
  Multiplex analyses of inflammatory markers (CRP)
1 month Postpartum Maternal Biomarkers (CRP) | 1 month postpartum
  Multiplex analyses of inflammatory markers (CRP)
6 month Postpartum Maternal Biomarkers (CRP) | 6 months postpartum
  Multiplex analyses of inflammatory markers (CRP)
12 month Postpartum Maternal Biomarkers (CRP) | 12 months postpartum
  Multiplex analyses of inflammatory markers (CRP)
16wk Maternal Biomarkers (IL6) | 16wks gestation
  Multiplex analyses of inflammatory markers (IL6)
36wk Maternal Biomarkers (IL6) | 36wks gestation
  Multiplex analyses of inflammatory markers (IL6)
1 month Postpartum Maternal Biomarkers (IL6) | 1 month postpartum
  Multiplex analyses of inflammatory markers (IL6)
6 month Postpartum Maternal Biomarkers (IL6) | 6 months postpartum
  Multiplex analyses of inflammatory markers (IL6)
12 month Postpartum Maternal Biomarkers (IL6) | 12 months postpartum
  Multiplex analyses of inflammatory markers (IL6)
16wks Maternal Biomarkers (adiponectin) | 16wks gestation
  Multiplex analyses of inflammatory markers (adiponectin)
36wks Maternal Biomarkers (adiponectin) | 36wks gestation
  Multiplex analyses of inflammatory markers (adiponectin)
1 month postpartum Maternal Biomarkers (adiponectin) | 1 month postpartum
  Multiplex analyses of inflammatory markers (adiponectin)
6 month postpartum Maternal Biomarkers (adiponectin) | 6 months postpartum
  Multiplex analyses of inflammatory markers (adiponectin)
12 month postpartum Maternal Biomarkers (adiponectin) | 12 months postpartum
  Multiplex analyses of inflammatory markers (adiponectin)
16wks Maternal Biomarkers (cortisol) | 16wks gestation
  Multiplex analyses of inflammatory markers (cortisol)
36wks Maternal Biomarkers (cortisol) | 36wks gestation
  Multiplex analyses of inflammatory markers (cortisol)
1 month Postpartum Maternal Biomarkers (cortisol) | 1 month postpartum
  Multiplex analyses of inflammatory markers (cortisol)
6 month Postpartum Maternal Biomarkers (cortisol) | 6 months postpartum
  Multiplex analyses of inflammatory markers (cortisol)
12 month Postpartum Maternal Biomarkers (cortisol) | 12 months postpartum
  Multiplex analyses of inflammatory markers (cortisol)

CONTACTS AND LOCATIONS:
Overall Officials: Linda May, MS, PhD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
de-identified data can be shared upon request to researchers